CLINICAL TRIAL: NCT01708408
Title: Measurement to Understand Reclassification of Disease of Cabarrus/Kannapolis The MURDOCK Study Registry and Biorepository Horizon 1.5
Brief Title: The MURDOCK Study Registry and Biorepository Horizon 1.5
Acronym: MURDOCK
Status: Active, not recruiting | Type: Observational
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00011196
Record Dates: First submitted 2012-10-15; First posted 2012-10-17 (Estimated); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Chronic Disease; Healthy Volunteers
Keywords: biorepository; biobank; registry; community; biospecimens; volunteers; chronic disease; longitudinal; blood; electronic health records; follow-up
MeSH Terms: conditions — Chronic Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, 25 mL (whole blood, plasma, serum, buffy coat, PAXgene); Urine, 36 mL
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- community
  Interventions: Genetic: Biomarker studies

INTERVENTIONS:
Genetic: Biomarker studies

SUMMARY:
The MURDOCK Study Community Registry and Biorepository (Horizon 1.5) aims to create a large-scale community registry and biorepository that can be used as a vehicle for future health services, epidemiologic, clinical trials and other omics-related research.

DETAILED DESCRIPTION:
The MURDOCK Study Community Registry and Biorepository's activities include enrolling approximately 50,000 participants who live in Cabarrus County and/or Kannapolis, North Carolina. Participants must consent to (1) use of the data provided by the participant through completion of the Participant Registry Questionnaire for epidemiologic population characterization, (2) annual contact to update their MURDOCK Horizon 1.5 database record, (3) release of their medical information, including but not limited to demographic information, problem lists, medications, social and family history, and results of laboratory and other testing modalities from pre-existing paper or electronic health records or electronic health records that may become available in the future, (4) provision of a blood and urine sample, and (5) contact up to four times/year to request participation in additional research studies.

ELIGIBILITY:
Inclusion Criteria:

1. A resident of Cabarrus County and/or the city of Kannapolis (and surrounding regions) for 6 or more months of the year
2. At least 18 years of age
3. Able to understand and give written informed consent, or have a legal guardian or caregiver present to give informed consent by proxy (assent from a participant between ages 12-18 will be obtained when their parent or legal guardian consents on their behalf).
4. Willing and able to participate in all 5 components of the registry and biorepository as described above in Section III

Exclusion Criteria:

1. There are no exclusions to participation if all inclusion criteria have been met.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The Community Registry and Biorepository is designed to create a community registry and biorepository populated by approximately 50,000 residents of Cabarrus County and/or the city of Kannapolis in North Carolina.
Sampling Method: Non-Probability Sample
Enrollment: 50000 (Estimated)
Dates: Start 2009-02 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
The MURDOCK Study Registry and Biorepository Horizon 1.5 | Upto 119 months
  To provide information for large-scale epidemiologic and clinical translational research and the research infrastructure to identify specific phenotypes and outcomes to improve medicine

CONTACTS AND LOCATIONS:
Overall Officials: Kristin M Newby, MD, Principal Investigator — Duke University
Locations (1):
- Duke Clinical Translational Science Institute-MURDOCK Study, Kannapolis, North Carolina, United States

REFERENCES:
- [Background] Tenenbaum JD, Christian V, Cornish MA, Dolor RJ, Dunham AA, Ginsburg GS, Kraus VB, McHutchison JG, Nahm ML, Newby LK, Svetkey LP, Udayakumar K, Califf RM. The MURDOCK Study: a long-term initiative for disease reclassification through advanced biomarker discovery and integration with electronic health records. Am J Transl Res. 2012;4(3):291-301. Epub 2012 Jul 23. PMID 22937207
- See also: MURDOCK Study website — http://www.murdock-study.org